CLINICAL TRIAL: NCT01327937
Title: A Prospective, Randomized, Controlled, Single-Site Post Marketing Study to Identify & Characterize the Molecular Mechanisms of Apligraf in Non-healing Wounds of Subjects With Venous Leg Ulcers
Brief Title: A Post Marketing Study of Apligraf in Non-healing Wounds of Subjects With Venous Leg Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 09-MOA-002-AG
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Venous Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apligraf Group (Active Comparator): Apligraf group - Applied at Day 0, Weeks 1-4 (maximum of 5 applications) Also cross-over at Week 4 for Control NPTH group - Apligraf applied at Week 4, Weeks 5-8 (maximum of 5 applications)
  Interventions: Device: Apligraf
- Standard of Care Dressing Group (Placebo Comparator): Standard of care dressing regimen - Foam dressing (eg, Mepilex) and 4 layered compression system (eg, Profore)
  Interventions: Other: Standard of Care Dressing Group

INTERVENTIONS:
Device: Apligraf — Apligraf group - Applied at Day 0, Weeks 1-4 (maximum of 5 applications) Also cross-over at Week 4 for Control NPTH group - Apligraf applied at Week 4, Weeks 5-8 (maximum of 5 applications)
  Arms: Apligraf Group
Other: Standard of Care Dressing Group — Standard dressing regimen - Foam dressing (eg, Mepilex) and 4 layered compression system (eg, Profore)
  Arms: Standard of Care Dressing Group

SUMMARY:
The overall study objective is to use microarray technology to identify and characterize the gene expression of multiple relevant genes in biopsies of non-healing venous ulcers.

DETAILED DESCRIPTION:
Subjects with a ≥5 cm2, non-infected target ulcer that has not reduced in area by ≥ 40% since the Screening visit will be randomized at Day 0 to either Apligraf or Control. After enrollment of 25 subjects, randomization will be discontinued and all remaining subjects will receive Apligraf.

Once the target ulcer is assessed by the Investigator as healed at a study visit, the subject's participation in the study is completed (eg, assessed as healed at Week 3, subject would not be required to complete any subsequent study visits).

Apligraf Group (Day 0 to Week 4) Prior to all applications, Apligraf will be fenestrated (perforated) in a standardized manner using a #11 blade with 6 fenestrations per 44 cm2.

For those subjects randomized to the Apligraf group, after Apligraf application, the dressing regimen will include a foam dressing (eg. Mepilex) and a 4 layered compression bandage system (eg. Profore) which will be changed weekly by the Investigator.

After the initial Apligraf application at study Day 0, Apligraf may be applied weekly thereafter for an additional 4 weeks at study Weeks 1, 2, 3, and 4, if, upon visual inspection, adherent Apligraf wound coverage is < 100%.

At Week 4, the area of the target ulcer will be compared to the area of the target ulcer at Day 0 to determine if the target ulcer is PTH or NPTH.

Apligraf subjects that do not achieve CWC by Week 5 will enter the Follow-Up Phase at that time.

Control Group (Day 0 to Week 4 [PTH] or Day 0 to Week 8 [NPTH] Beginning at Day 0, subjects randomized to the Control group will receive the standard dressing regimen which includes a foam dressing (e.g. Mepilex®) and a four layered compression bandage system (e.g. Profore™) which will be changed weekly by the Investigator.

At study Week 4, the size of the ulcer will be compared to the size at study Day 0 to determine if the ulcer is demonstrating "Predicted to Heal" (PTH), defined as >40% reduction in ulcer surface area compared with study Day 0, or "Not Predicted to Heal (NPTH), defined as <40% reduction in ulcer surface area compared with study Day 0.

Control PTH subjects that do not achieve CWC by Week 4 will continue to receive Control treatment and will enter the Follow-Up Phase at Week 5.

Control NPTH subjects will receive Apligraf beginning at Week 4. Prior to all applications, Apligraf will be fenestrated (perforated) in a standardized manner using a #11 blade with 6 fenestrations per 44 cm2. After the initial Apligraf application at Week 4, Apligraf may be applied weekly thereafter for an additional 4 weeks at study Weeks 5, 6, 7, and 8 if upon visual inspection, adherent Apligraf wound coverage is < 100%. After Apligraf application, the standard dressing regimen will be applied over the target ulcer. The dressing will be changed weekly by the Investigator. At Week 8, the area of the target ulcer will be compared to the area of the target ulcer at Week 4 to determine if the target ulcer is PTH or NPTH.

Control NPTH subjects that do not achieve CWC by Week 9 will enter the Follow-up Phase at that time.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has at least 1 clinically non-infected full-thickness venous leg ulcer (VLU) at least 5 cm2 in size.
2. Subject is at least 18 years of age or older.
3. Subject must have read, understood and signed an institutional review board (IRB) approved Informed Consent Form.
4. Subject must be able and willing to follow study procedures and instructions.

Exclusion Criteria:

1. Subjects who require VAC® (Vacuum Assisted Closure™) therapy on or after Day 0 Study visit.
2. Subject has arterial disease as determined by an Ankle Brachial Index (ABI) measurement of <0.65.
3. Subject with any systemic or congenital condition like uncontrolled diabetes mellitus, positive HIV test, or any disorder(s) that may compromise wound healing.
4. Subjects with carcinomas located at the target ulcer with biopsy confirmed active malignancy. (Subjects with other carcinoma locations would not be excluded from entry into the study.)
5. Subjects who are currently receiving, or have received at any time within 30 days prior to Screening visit, non-inhaled corticosteroids except topical steroids not at the target ulcer (Inhaled steroid therapy is acceptable on study.), immunosuppressive agents, radiation therapy, hemodialysis, peritoneal dialysis or chemotherapy. (Anticipated use of the above agents or therapies would exclude subject from entry into the study.)
6. Clinical vasculitis, severe rheumatoid arthritis, and other collagen vascular diseases.
7. Signs and symptoms of cellulitis or osteomyelitis at the target ulcer.
8. Avascular target ulcer beds. (Ulcers of mixed etiology such as arterial disease with VLU will be excluded.)
9. Target ulcer with exposed bone, tendon or fascia.
10. Known hypersensitivity to bovine collagen or to the components of the Apligraf agarose shipping medium.
11. Subject enrolled in any wound or investigational study (drug, biologic or device) for any disease within 30 days of the Screening visit.
12. Subject previously treated with Apligraf, Dermagraft® or any other cell therapy at the target ulcer site within 30 days of the Screening visit.
13. Subject with a history of alcohol or substance abuse within the previous year, which could interfere with study compliance such as inability to attend scheduled study visits.
14. Subject who is a current smoker or has not ceased smoking 6 months prior to the Screening visit, or in the opinion of the Investigator, has a smoking history that may compromise wound healing.
15. Subject who, in the opinion of the Investigator, for any reason other than those listed above, will not be able to complete the study per protocol.
16. Target ulcer has not decreased in size by > 40% from Screening to Day 0.
17. Confirmed gene expression overlap between the subject's cells (buccal swab) and the cells contained in Apligraf.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Determine changes in gene expression in subjects receiving Apligraf (includes Apligraf & Control NPTH) compared to 1 week post treatment | Apligraf group - Day 0 & Week 1; Control NPTH group-Weeks 4 & 5
  Not Predicted to Heal (NPTH) defined as <40% reduction in ulcer surface area from Day 0 to Week 4

SECONDARY OUTCOMES:
Determine changes in gene expression in subjects receiving Apligraf (includes Apligraf & Control NPTH)compared to subjects not receiving Apligraf at time of initial treatment and at 1 week post treatment | Apligraf group-Day 0 & Week 1; Control NPTH group-Weeks 4 & 5
  NPTH defined as above
Determine differences in gene expression in following groups (see description section) | Apligraf group-Day 0 & Week 1; Control NPTH group-Weeks 4 & 5
  1. Apligraf (APG) subjects Predicted to Heal (PTH) compared to Apligraf subjects Not Predicted to Heal (NPTH)
  2. APG subjects PTH compared to Control subjects PTH
  3. APG subjects NPTH compared to Control subjects NPTH
  4. Control subjects PTH compared to Control subjects NPTH
  5. All subjects (Apligraf and Control) PTH compared to all subjects NPTH
  Also evaluate validity of surrogate endpoint (ulcer decrease of>/= 40% from Day 0 to Week 4) for complete wound closure (CWC*) by Week 24
  * CWC defined as 100% epithelialization with absence of drainage

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Badiavas, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Stone RC, Stojadinovic O, Sawaya AP, Glinos GD, Lindley LE, Pastar I, Badiavas E, Tomic-Canic M. A bioengineered living cell construct activates metallothionein/zinc/MMP8 and inhibits TGFbeta to stimulate remodeling of fibrotic venous leg ulcers. Wound Repair Regen. 2020 Mar;28(2):164-176. doi: 10.1111/wrr.12778. Epub 2019 Dec 4. PMID 31674093
- [Derived] Stone RC, Stojadinovic O, Rosa AM, Ramirez HA, Badiavas E, Blumenberg M, Tomic-Canic M. A bioengineered living cell construct activates an acute wound healing response in venous leg ulcers. Sci Transl Med. 2017 Jan 4;9(371):eaaf8611. doi: 10.1126/scitranslmed.aaf8611. PMID 28053158